CLINICAL TRIAL: NCT05055102
Title: Post-Market Clinical Follow-up of WOVEX (Wovex® Polyester Vascular Prostheses) Bifurcated Prostheses From LEMAITRE VASCULAR Society in the Treatment of Aneurysms or Occlusive Diseases of the Abdominal Aorta
Acronym: WOBIF
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: STEINMETZ LEMAITRE 2020
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Aneurysms or Occlusive Disease of the Abdominal Aorta
MeSH Terms: conditions — Aneurysm | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with WOVEX bifurcated prosthesis: * Patients who have undergone open abdominal aortic surgery between January 1st, 2013 and December 31, 2017 in Burgundy Dijon Hospital.
  * Patients who have been treated with a WOVEX bifurcated prosthesis (Wovex® Polyester Vascular Protheses)
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — demographics co-morbidities risk factors operative, hospital and vascular follow-up data

SUMMARY:
The Wovex bifurcated dacron vascular prostheses have been available on the French market since 2008. They are mainly used to treat aneurysmal or occlusive aortic diseases. To date, they have not been the subject of a specific clinical efficacy/safety study, unlike other Dacron prostheses used in the same field.

We purpose a monocentric, retrospective, consecutive study based on medical data, including all the patients operated for aneurysms or occlusive disease of the abdominal aorta at Dijon Bourgogne University Hospital between 2013 and 2017 and who received a WOVEX bifurcated prosthesis (Wovex® Polyester Vascular Protheses).

The objective is to explore the safety (short-term postoperative morbidity and mortality at 5 years) and efficacy (primary permeability, secondary permeability and dilatation of the prosthesis at 5 years) of the WOVEX prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is volontarily agree to participation
* Patients operated for aneurysms or occlusive disease of the abdominal aorta at Dijon Bourgogne University Hospital between January, 1st 2013 and December 31, 2017 who received a WOVEX bifurcated prosthesis (Wovex® Polyester Vascular Protheses) from LEMAITRE VASCULAR Society

Exclusion Criteria:

- Deceased patients who have expressed their refusal of post-mortem processing of their personal health data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated for aneurysms or occlusive disease of the abdominal aorta at Dijon Bourgogne University Hospital between January, 1st 2013 and December 31, 2017 who received a WOVEX bifurcated prosthesis (Wovex® Polyester Vascular Protheses) from LEMAITRE VASCULAR Society
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2021-01-16 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Safety and security | 5 years
  Occurrence of death or major re-intervention (bypass stenosis/thrombosis, false anastomotic aneurysm, prosthesis infection, anastomosis rupture, amputation) over the entire follow-up period (from date of surgery to study end date (February 28, 2021))

SECONDARY OUTCOMES:
Major surgical reintervention | 5 years
  bypass stenosis/thrombosis, false anastomotic aneurysm, prosthesis infection, anastomosis rupture, amputation throughout the follow-up period
Primary permeability | 5 years
  Stenosis/thrombosis of the prosthesis over the entire follow-up period
Secondary permeability | 5 years
  Stenosis/thrombosis after reintervention over the entire follow-up period
Dilatation of the prothesis | 5 years
  Diameter of the prosthesis over the entire follow-up period
Occurence of MAVE and MACE | 5 years
  Occurence of MAVE and MACCE (re-interventions, ischemic cardiac, neurological (stroke/TIA), pulmonary and renal complications) throughout the follow-up period
Occurence of adverse events | 5 years
  Other adverse events over the entire follox-up period

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France